CLINICAL TRIAL: NCT04882969
Title: A Pilot Study Evaluating the Safety and Efficacy of a Fractionated Thulium Laser and KeraFactor for the Treatment of Alopecia
Brief Title: Thulium Laser and KeraFactor for the Treatment of Androgenetic Alopecia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed Indication
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Kseniya Kobets, Assistant Professor, Department of Medicine (Dermatology), Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12914
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Androgenetic Alopecia
Keywords: alopecia; androgenetic; laser; hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Each participating subject will serve as his or her baseline control and will receive up to two (2) treatments per month for 3 months with Thulium laser and post-laser treatment topically applied Kerafactor.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fractionated Thulium Laser and KeraFactor (Experimental): All participating subjects will serve as their own baseline control and will receive treatment of their androgenetic alopecia with LaseMD, a 1927nm Fractionated Thulium laser and post-treatment topically applied KeraFactor every 2 weeks for 12 week period.
  Interventions: Device: Fractionated Thulium laser

INTERVENTIONS:
Device: Fractionated Thulium laser — LaseMD Lutronic Laser is a 1927-nm fractionated thulium laser, which is better absorbed by water than non-ablative 1,540-nm erbium glass laser energy. The laser energy and power can be customized to target a specific penetration depth and achieve selective photothermolysis in skin while mitigating injury to surrounding tissue. The thermal energy generated by the laser has been shown to facilitate the delivery of kerafactor, which contain hair growth factors to stimulate follicular progenitor cell proliferation and differentiation into follicular keratinocytes to promote hair growth.
  Other Names: LaseMD Lutronic Laser

SUMMARY:
The objective of this clinical study is to assess the safety and efficacy of using a laser and hair growth factors in the treatment of male-pattern hair loss. Participating subjects will receive up to two (2) treatments per month for 6 months with the laser and post-treatment topically applied hair growth factors and will have a 6 month follow-up period.

DETAILED DESCRIPTION:
This is a single-center, open-label, baseline-controlled, study evaluating the use of a Thulium laser (1927nm) and post-treatment topically applied KeraFactor, which contain hair-stimulating growth factors, in the treatment of androgenetic alopecia. The study may enroll up to 20 subjects looking for improvement in their hair loss. Multiple treatment areas per subject may be included. Each subject will receive up to two (2) treatments per month over a 3-month period. Follow Up Visits are planned for 3, and 9 months post last treatment. Standardized photography of the treatment areas will be recorded Pre and Post Treatment at each visit. Measurement outcomes will be compared to baseline. During the initial visit, subjects who meet the study's eligibility criteria will receive the first treatment after signing informed consent form.

The follow up phase will consist of before and after photographs graded by blinded observers. Subjects are instructed to inform clinical staff after the treatment if they experience any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and date an IRB approved informed consent form
* Subjects with diagnosis of androgenetic alopecia with hair loss recorded over the past 6 months. (Ludwig Savin Scale: Class I-4, II-1, II-2 for females and Norwood Hamilton Class 3-4 for males
* Able to read, understand and voluntarily provide written informed consent.
* Healthy male or female, ≥ 18 years of age at time of informed consent up to 65 years of age, seeking treatment for hair loss.
* Subject is determined to be healthy, non-smoker who agrees not to make any changes to their daily hair treatment regime during the study.
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Women of child-bearing age are required to be using a reliable, non-hormonal method of birth control for the duration of the study. Subjects will be asked to have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

* Subjects does not have the capacity to consent to the study
* Subject has other types of alopecia of the scalp (i.g., alopecia areata, scarring alopecia)
* Use of minoxidil or 5-alpha reductase inhibitors (i.e., finasteride, dutasteride) 3 months prior to screening date.
* Any medical condition that in the consideration of the investigator, would present an increased risk of a photosensitivity reaction to the subject.
* Pregnant in the last 12 months, intending to become pregnant, postpartum or nursing in the last 12 months.
* Any previous surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months.
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy for prior 12 months.
* History or current use of the following prescription medications: Immunosuppressive medications/biologics, 6 months prior to and during the study. Accutane or other systemic retinoids within the past twelve months.
* Smoking or vaping in the past 12 months.
* History of hyperlipidemia, diabetes mellitus, hepatitis, or bleeding disorders.
* History of major depressive disorders or endocrine disorders including but not limited to; hypothyroidism, Hashimoto's thyroiditis, or hyperthyroidism as well as Polycystic Ovarian Syndrome (PCOS) in females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with score of 2 or 3 on Clinician Global Aesthetic Improvement (CGAIS) scale at week 12 of treatment. | 12 weeks
  Clinician Global Aesthetic Improvement Scale (CGAIS) is a Likert scale, ranging from "greatly decreased (-3)" hair growth to "greatly increased (+3)" hair growth.
  1. Greatly decreased (-3)
  2. Moderately decreased (-2)
  3. Slightly decreased (-1)
  4. No change (0)
  5. Slightly increased (+1)
  6. Moderately increased (+2)
  7. Greatly increased (+3)
  Based on a live assessment of the subject while referring to the subject's pre-treatment scalp photographs, the clinician will make an assessment of post-treatment hair growth.
Percentage of subjects with score of 2 or 3 on Subject Global Aesthetic Improvement at week 12 of treatment. | 12 weeks
  Subject Global Aesthetic Improvement Scale (SGAIS) is a Likert scale, ranging from "greatly decreased (-3)" hair growth to "greatly increased (+3)" hair growth.
  1. Greatly decreased (-3)
  2. Moderately decreased (-2)
  3. Slightly decreased (-1)
  4. No change (0)
  5. Slightly increased (+1)
  6. Moderately increased (+2)
  7. Greatly increased (+3)
  Subjects will be given a hand mirror for self-assessment of post-treatment hair growth compared to subject's pre-treatment scalp photographs.

SECONDARY OUTCOMES:
Percentage of subjects with score of 2 or 3 on Patient Satisfaction Questionnaire at week 12 of treatment. | 12 weeks
  Patient Satisfaction Questionnaire will use Lickert scale, ranging from "greatly decreased (-3)" to "greatly increased (+3)".
  1. Greatly decreased (-3)
  2. Moderately decreased (-2)
  3. Slightly decreased (-1)
  4. No change (0)
  5. Slightly increased (+1)
  6. Moderately increased (+2)
  7. Greatly increased (+3)
  The seven point Lickert scale will apply to following patient satisfaction questions:
  1. Please choose the option that better represents the change in how your hair looks OVERALL in the area treated?
  2. Please choose the option that better represents the change in your hair THICKNESS in the area treated?
  3. Please choose the option that better represents the change in your hair SHEDDING/LOSS in the area treated?
  4. Please choose the option that better represents the change in your hair DARKNESS in the area treated.
Reported pain score on Numeric Rating Scale for Pain | 12 weeks
  The Numeric Rating Scale for Pain is an 11-point scale scored from 0-10, with 0 = no pain, 5 = moderate pain, and 10 = worst possible pain. Subjects select a value that is most in line with the intensity of their pain experienced during and after treatment with Thulium Laser and topical Kerafactor.

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States